CLINICAL TRIAL: NCT06282627
Title: Prospective Cohort Study of Non-hospitalised COVID-19 Patients: Determining Length of Isolation and Patient Clinical Development at Home (COVID-HOME Study)
Brief Title: The COVID HOME Study: Prospective Cohort Study of Non-hospitalised COVID-19 Patients
Acronym: COVID-HOME
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 10430012010023
Record Dates: First submitted 2024-02-26; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Post-COVID-19 Syndrome
Keywords: COVID-19; SARS-CoV-2; Non-hospitalised; Post-COVID-19 Syndrome
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-hospitalised individuals: No intervention. Observational study
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — No intervention. Observational study

SUMMARY:
Background. Guidelines on COVID-19 management are developed as we learn from this pandemic. However, most research has been done on hospitalised patients and the impact of the disease on non-hospitalised and their role in transmission are not yet well understood.

The COVID HOME study conducts research among COVID-19 patients and their family members who were not hospitalised during acute disease, to guide patient care and inform public health guidelines for infection prevention and control in the community and household.

Methods. An ongoing prospective longitudinal observational study of COVID-19 outpatients was established in March 2020 at the beginning of the COVID-19 pandemic in the Netherlands. Laboratory confirmed SARS-CoV-2 infected individuals of all ages that did not merit hospitalisation, and their household (HH) members, were enrolled after written informed consent. Enrolled participants were visited at home within 48 hours after initial diagnosis, and then weekly on days 7, 14 and 21 to obtain clinical data, a blood sample for biochemical parameters/cytokines and serological determination; and a nasopharyngeal/throat swab plus urine, stool and sperm or vaginal secretion (if consenting) to test for SARS-CoV-2 by RT-PCR (viral shedding) and for viral culturing. Weekly nasopharyngeal/throat swabs and stool samples, plus a blood sample on days 0 and 21 were also taken from HH members to determine whether and when they became infected. All participants were invited to continue follow-up at 3-, 6-, 12- and 18-months post-infection to assess long-term sequelae and immunological status.

DETAILED DESCRIPTION:
An ongoing prospective longitudinal observational study of SARS-CoV-2 infected individuals that did not require hospitalisation and their HH members was initiated on March 2020, at the start of the pandemic in the Netherlands.

Enrolled individuals comprised the identified laboratory COVID-19 index positive patients plus all their HH members. The average number of HH inhabitants in the Netherlands and the northern region is 2.14 [44], thus for each enrolled patient we expected to enrol an average of 1-2 HH members in addition. Patients were followed daily at home approximately during 3 weeks post-infection to characterize their acute clinical phenotype, and are currently being followed at 3, 6, 12 and 18 months to determine their long-term clinical and serological evolution. During the follow-up, clinical data and different types of samples were/are collected, as described below.

ELIGIBILITY:
Inclusion Criteria:

* Onset of symptoms <5 days before inclusion
* Positive diagnostic RT-PCR for SARS-CoV-2 performed within 48h of inclusion
* Index person should supply all required samples in the protocol for the duration of the study
* All HH members should join the study
* Signing of informed consent form

Exclusion Criteria:

* False positive RT-PCR test
* Non compliance with study follow-up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study is carried out amongst residents of the Northern Provinces of the Netherlands (Groningen, Friesland, Overijssel and Drenthe) comprising around 1.7 million inhabitants. Laboratory confirmed SARS-CoV-2 infected individuals of all ages (index cases) that do not merit hospitalisation, and their HH members, were invited to join the study and enrolled after signing a written informed consent. Consenting parents/guardians of infected children (≤16 years) signed the informed consent form. The complete HH, i.e. all persons (contacts) living in the same home, was to join the study at enrolment. If this requirement was not fulfilled, the HH was excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infection | Three weeks of acute follow-up
  SARS-CoV-2 positive individuals by qRT-PCR

SECONDARY OUTCOMES:
Long-term sequelae | 2 years
  Reporting at least one symptom at 3, 6, 12 months post-infection

CONTACTS AND LOCATIONS:
Overall Officials: Adriana TAMI, Principal Investigator — University Medical Center Groningen, University of Groningen, Groningen, The Netherlads
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Tami A, van der Gun BTF, Wold KI, Vincenti-Gonzalez MF, Veloo ACM, Knoester M, Harmsma VPR, de Boer GC, Huckriede ALW, Pantano D, Gard L, Rodenhuis-Zybert IA, Upasani V, Smit J, Dijkstra AE, de Haan JJ, van Elst JM, van den Boogaard J, O' Boyle S, Nacul L, Niesters HGM, Friedrich AW. The COVID HOME study research protocol: Prospective cohort study of non-hospitalised COVID-19 patients. PLoS One. 2022 Nov 3;17(11):e0273599. doi: 10.1371/journal.pone.0273599. eCollection 2022. PMID 36327223
- See also: Study protocol — https://doi.org/10.1371/journal.pone.0273599